CLINICAL TRIAL: NCT03959254
Title: EFFECTIVENESS OF A PROTOCOLIZED TREATMENT OF SPECIFIC PHYSIOTHERAPY FOR SUBJECTS SURGICALLY OPERATED BY ARTHROSCOPY FOR FEMOROACETABULAR SYNDROME
Brief Title: Specific Protocoled Physiotherapy Treatment for Subjects Surgically Treated for Femoroacetabular Syndrome
Acronym: FAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU UCH FAI
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Application of a protocol of active exercises for recovery after arthroscopic hip surgery, adapted to the femoroacetabular shock characteristics.
  Interventions: Procedure: Physiotherapy post-surgical protocol for femoroacetabular impingement
- Control Group (Active Comparator): Usual post-surgical general guidelines for hip interventions described by Gocen et al
  Interventions: Procedure: Physiotherapy post-surgical protocol for femoroacetabular impingement

INTERVENTIONS:
Procedure: Physiotherapy post-surgical protocol for femoroacetabular impingement — The intervention is structured in 14 weeks. Gradually the level of demand for the exercises increases over the weeks. Isometric and concentric exercises of the affected muscle groups are combined in the first weeks, as well as mobilization exercises of the joints involved in the injury. In addition, the time of permanence in a sitting, prone or supine position is prescribed. The return to the march and activities of daily life are staggered.
  The number of series and repetitions to be performed is described in each exercise.

SUMMARY:
Physiotherapy treatment protocols described in the bibliography after hip surgery are most of them nonspecific. An experimental study is proposed to determine the effectiveness of a protocolized treatment of physiotherapy in the postoperative treatment of femoroacetabular impingement treated by arthroscopy. This study tries to adapt the non-specific post-surgical physiotherapy treatment protocols of the hip to the characteristics of the femoroacetabular impingement and its arthroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered hip / groin pain for at least 3 months.
* Be a patient diagnosed with femoroacetabular syndrome by an orthopedic surgeon based on symptoms, clinical signs and diagnostic imaging.
* To have signed the informed consent.
* Have time available to follow a 14-week physiotherapy treatment program.
* Be programmed for hip arthroscopy.
* Be able to speak and understand the Spanish language.
* Be between 18 and 50 years of age.

Exclusion Criteria:

* To have received physiotherapy treatment in the last three months.
* Having previously received hip surgery.
* Subjects with previous deformities in the femur that severely alter joint mobility such as Perthes disease, gliding of the upper femoral epiphysis or avascular necrosis, acetabular fracture, hip dislocation or fracture of the femoral neck.
* Evidence of preexisting osteoarthritis, defined as Tonnis grade> 2
* Subjects with previous deformities in the pelvis that severely alter joint mobility.
* Any other cardiovascular, psychological and / or cognitive diagnosed pathology that impedes the correct understanding of the study and prevents objective study variables.
* Subjects that are under the effects of anesthetics or muscle relaxants that mask the sensation of the patient before the techniques of the study.
* Professional athletes.
* Subjects in which hip arthroscopy is contraindicated.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Hip Range of Mobility | 14 weeks
  The range of mobility is evaluated by goniometry.
Intensity of pain | 14 weeks
  The intensity of pain is evaluated by Visual Analogue Scale (VAS). The values are between 0 (absence of pain) to 10 (maximum intensity pain)
Functionality of the hip | 14 weeks
  Modified Harris Hip Score Questionnaire (mHHS) is used to determine the functionality of the hip. The values are between 0 (lowest functionality) and 100 (normal function). The sub scales the subscales that compose it are hip pain (from 0 to 44), lameness in walking (from 0 to 11), need for walking aids (0 to 11), walked distance (0 to 11), ability to going up or down stairs (0 to 4), putting on shoes (0 to 4), sitting down without pain (0 to 5) and possibility of using public transport (0 to 1), with 0 being always the worst value.
Fabere Test | 14 weeks
  The patient's hip is flexed, abducted and externally rotated by placing the external malleolus on the knee of the contralateral leg. The pelvis is stabilized and an overpressure is applied to the inside of the knee. It is positive if the pain in the buttock or groin is reproduced. Test with inter-evaluator reliability in Kappa values (95% CI) of 0.60
Faddir Test | 14 weeks
  Flexion, adduction and internal rotation test. The supine patient, the evaluator patiently brings the patient's hip up to 100º flexion and adduction while applying internal rotation. It is positive if pain in the groin is reproduced. Test with inter-evaluator reliability in Kappa values of 0.48
Ober test | 14 weeks
  Patient in lateral decubitus position. The evaluator flexes the knee that is evaluated at 90º and abducts and extends the hip until it is level with the trunk. The evaluator lets the gravity bring the hip on aduction as possible. Test with inter-evaluator reliability of 0.90

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad CEU Cardenal Herrera, Valencia, Moncada
  - Ceu Cardenal Herrera University, Moncada, Valencia

REFERENCES:
- [Background] Smith-Petersen MN. The classic: Treatment of malum coxae senilis, old slipped upper femoral epiphysis, intrapelvic protrusion of the acetabulum, and coxa plana by means of acetabuloplasty. 1936. Clin Orthop Relat Res. 2009 Mar;467(3):608-15. doi: 10.1007/s11999-008-0670-0. Epub 2008 Dec 17. PMID 19089521
- [Background] Leunig M, Podeszwa D, Beck M, Werlen S, Ganz R. Magnetic resonance arthrography of labral disorders in hips with dysplasia and impingement. Clin Orthop Relat Res. 2004 Jan;(418):74-80. doi: 10.1097/00003086-200401000-00013. PMID 15043096
- [Background] Griffin DR, Dickenson EJ, Wall PDH, Achana F, Donovan JL, Griffin J, Hobson R, Hutchinson CE, Jepson M, Parsons NR, Petrou S, Realpe A, Smith J, Foster NE; FASHIoN Study Group. Hip arthroscopy versus best conservative care for the treatment of femoroacetabular impingement syndrome (UK FASHIoN): a multicentre randomised controlled trial. Lancet. 2018 Jun 2;391(10136):2225-2235. doi: 10.1016/S0140-6736(18)31202-9. Epub 2018 Jun 1. PMID 29893223
- [Background] Kuhns BD, Weber AE, Batko B, Nho SJ, Stegemann C. A FOUR-PHASE PHYSICAL THERAPY REGIMEN FOR RETURNING ATHLETES TO SPORT FOLLOWING HIP ARTHROSCOPY FOR FEMOROACETABULAR IMPINGEMENT WITH ROUTINE CAPSULAR CLOSURE. Int J Sports Phys Ther. 2017 Aug;12(4):683-696. PMID 28900574
- [Background] Wall PD, Dickenson EJ, Robinson D, Hughes I, Realpe A, Hobson R, Griffin DR, Foster NE. Personalised Hip Therapy: development of a non-operative protocol to treat femoroacetabular impingement syndrome in the FASHIoN randomised controlled trial. Br J Sports Med. 2016 Oct;50(19):1217-23. doi: 10.1136/bjsports-2016-096368. PMID 27629405
- [Background] Bennell KL, O'Donnell JM, Takla A, Spiers LN, Hunter DJ, Staples M, Hinman RS. Efficacy of a physiotherapy rehabilitation program for individuals undergoing arthroscopic management of femoroacetabular impingement - the FAIR trial: a randomised controlled trial protocol. BMC Musculoskelet Disord. 2014 Feb 26;15:58. doi: 10.1186/1471-2474-15-58. PMID 24571824
- [Background] Gocen Z, Sen A, Unver B, Karatosun V, Gunal I. The effect of preoperative physiotherapy and education on the outcome of total hip replacement: a prospective randomized controlled trial. Clin Rehabil. 2004 Jun;18(4):353-8. doi: 10.1191/0269215504cr758oa. PMID 15180117
- [Background] Kemp JL, Coburn SL, Jones DM, Crossley KM. The Physiotherapy for Femoroacetabular Impingement Rehabilitation STudy (physioFIRST): A Pilot Randomized Controlled Trial. J Orthop Sports Phys Ther. 2018 Apr;48(4):307-315. doi: 10.2519/jospt.2018.7941. PMID 29607766
- See also: The University CEU-Cardenal Herrera is the first private university in the Valencian Community. It belongs to the Foundation San Pablo CEU, the leading educational organization in Spain with three Universities all over Spain. — http://www.uchceu.es

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03959254/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03959254/ICF_001.pdf